CLINICAL TRIAL: NCT04250155
Title: A Phase Ia/Ib, Open-Label, Multicenter, Global, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of XmAb24306 as a Single Agent and in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: An Open-Label Dose-Escalation Study to Evaluate XmAb24306 as a Single Agent and in Combination With Atezolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO41596
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a Dose Escalation (Experimental): Participants will receive XmAb24306 until study treatment discontinuation or study termination.
  Interventions: Drug: XmAb24306
- Phase 1a Dose Expansion (Experimental): Participants will receive XmAb24306 until study treatment discontinuation or study termination.
  Interventions: Drug: XmAb24306
- Phase 1b Dose Escalation (Experimental): Participants will receive XmAb24306 and atezolizumab until study treatment discontinuation or study termination.
  Interventions: Drug: Atezolizumab; Drug: XmAb24306
- Phase 1b Dose Expansion (Experimental): Participants will receive XmAb24306 and atezolizumab until study treatment discontinuation or study termination.
  Interventions: Drug: Atezolizumab; Drug: XmAb24306

INTERVENTIONS:
Drug: XmAb24306 — Participants will receive intravenous (IV) XmAb24306.
  Other Names: RO7310729
  Arms: Phase 1a Dose Escalation; Phase 1a Dose Expansion
Drug: Atezolizumab — Participants will receive IV XmAb24306 followed by IV atezolizumab
  Other Names: RO5541267
  Arms: Phase 1b Dose Escalation; Phase 1b Dose Expansion
Drug: XmAb24306 — Participants will receive IV XmAb24306 followed by IV atezolizumab.
  Other Names: RO7310729
  Arms: Phase 1b Dose Escalation; Phase 1b Dose Expansion

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and activity of XmAb24306 alone or in combination with a checkpoint inhibitor treatment in participants with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Key General Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >/= 12 weeks
* Adequate hematologic and end-organ function
* For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative serum pregnancy test for women of childbearing potential
* Histologically confirmed locally advanced, recurrent, or metastatic incurable solid tumor malignancy
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Availability of representative tumor specimens

Key General Exclusion Criteria

* Pregnant or breastfeeding, or intending to become pregnant during the study
* Significant cardiovascular disease
* Current treatment with medications that prolong the QT interval
* Known clinically significant liver disease
* Poorly controlled Type 2 diabetes mellitus
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* History of malignancy other than disease under study within 3 years prior to screening
* Active or history of autoimmune disease or immune deficiency
* Active tuberculosis, hepatitis B, hepatitis C, or known/suspected Epstein Barr virus infection
* Positive for HIV infection
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to approximately 4 years

SECONDARY OUTCOMES:
Serum Concentration of XmAb24306 | Baseline, then at pre-defined intervals for the first year of treatment or until participant discontinues study treatment
Objective Response Rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 4 years
Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1 | Up to approximately 4 years
Progression-Free Survival (PFS) as Determined by the Investigator According to RECIST v1.1 | Up to approximately 4 years
ORR as Based on Radiographic Assessment by the Investigator Using Modified RECIST v1.1 for Immune-Based Therapeutics (iRECIST) | Up to approximately 4 years
DOR as Based on Radiographic Assessment by the Investigator Using iRECIST | Up to approximately 4 years
PFS as Based on Radiographic Assessment by the Investigator Using iRECIST | Up to approximately 4 years
Overall Survival (OS) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (6):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Stanford Health Centre - Palo Alto, Palo Alto, California
  - University of California, San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale University, New Haven, Connecticut
  - City of Hope Comprehensive Cancer Center, Ann Arbor, Michigan
  - SCRI Oncology Partners, Nashville, Tennessee
- Parkville Cancer Clinical Trial Unit (PCCTU), Melbourne, Victoria, Australia
- GasthuisZusters Antwerpen, Wilrijk, Antwerp, Belgium
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
- Netherlands (2):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen, Groningen
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (5):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Cordoba
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra-Madrid, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing